CLINICAL TRIAL: NCT06268639
Title: Evaluation of Bone Density Before and After Placement of Implant Using Osseodensification Technique
Acronym: BIDOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Assistant Professor, King Khalid University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECM#2024-216; RGP1/347/44 (Other Grant/Funding Number: King Khalid University)
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Evaluation of Osseointegration and Stability of Dental Implants in Bone Density Enhanced by Osseodensification Technique
Keywords: Osseodensification; Dental implants; Bone density; Primary stability; Osteotomy

STUDY DESIGN:
Intervention Model Description: The study employs a single-group, interventional model to examine the impact of osseodensification on bone density at dental implant sites. It involves a sequential process starting from pre-operative bone density assessment using DentaScan CT, followed by surgical intervention using osseodensification drills, and concluding with a post-operative bone density evaluation to compare changes. This approach aims to determine if osseodensification can significantly enhance bone density and stability around implant sites, thereby potentially improving the success rates of dental implants. The methodology includes detailed pre-operative and post-operative assessments, with statistical analysis conducted to evaluate the effectiveness of the intervention.
Masking Description: The study employs an open-label design, where no masking is applied. This means that the participants, care providers, investigators, and outcomes assessors are all aware of the intervention being administered. Given the nature of the intervention-osseodensification technique used in dental implant surgery-it is not feasible to blind the study participants or the clinical staff involved in the procedure and assessment to the intervention being studied. The open-label approach allows for direct observation of the intervention's effects on bone density without the complexity of blinding, which is often the case in surgical and procedural interventions where the treatment administered is evident.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osseodensification in Dental Implant Surgery (Experimental): The arm involves participants undergoing dental implant surgery with the use of osseodensification drills. This technique is intended to enhance bone density and improve the primary stability of the implants by compacting bone rather than removing it during the osteotomy process. The study aims to assess the impact of osseodensification on bone density at the implant sites, comparing pre-operative and post-operative bone density measurements to evaluate the effectiveness of this intervention.
  Interventions: Procedure: Osseodensification

INTERVENTIONS:
Procedure: Osseodensification — The intervention, osseodensification, involves a surgical technique using specific drills (e.g., Densah burs) rotated in a counterclockwise direction to compact bone rather than remove it, thereby increasing bone density around the implant site. This method is aimed at improving the primary stability of dental implants by creating a denser bone environment, which theoretically should lead to better osseointegration and long-term success of the implant. The technique distinguishes itself from traditional drilling by preserving and enhancing bone structure, which is crucial for the success of dental implants in patients.

SUMMARY:
The study investigates the impact of osseodensification drills on bone density changes surrounding dental implants. Osseodensification, a novel technique, is hypothesized to enhance primary stability of implants by densifying bone rather than removing it during osteotomy. Participants undergo pre-operative and post-operative DentaScan CT analyses to measure bone density in Hounsfield units at apical, mesial, and distal positions around the implant sites. This intervention-based research aims to quantify the benefits of osseodensification in improving bone quality and implant success. Data from 32 sites, analyzed via the Radiant DICOM software, undergo statistical examination using SPSS to ascertain significant differences in bone density pre- and post-surgery. The outcome could redefine surgical approaches in implantology, emphasizing osseodensification's role in achieving superior bone-implant integration.

DETAILED DESCRIPTION:
Study Design The research is an interventional study targeting a single group of patients slated for dental implant placement, incorporating a total of 32 implant sites for detailed analysis. The study is meticulously designed to track each participant through sequential phases, including pre-operative evaluation, the surgical intervention employing osseodensification drills, and a thorough post-operative assessment to gauge the technique's impact on bone density and implant stability.

Pre-operative Evaluation Participants undergo a comprehensive dental examination before the surgical procedure, which includes DentaScan CT imaging conducted at Rohilkhand Medical College and Hospital's Department of Radiology. The imaging, analyzed using Radiant DICOM software, facilitates precise measurement of bone density at strategic locations around the planned implant sites, specifically at apical, mesial, and distal positions. These measurements, recorded in Hounsfield units, establish baseline bone density values for each site, grouped as Group 1 for analysis.

Surgical Procedure Implant placement surgeries are carried out under local anesthesia in the Department of Prosthodontics. Initial osteotomy sites are prepared using a pilot drill, followed by the application of osseodensification drills (VT1525 and VT2535) in a non-cutting, counterclockwise direction to expand and densify the bone at the osteotomy sites. This technique is theorized to enhance primary stability of the implants by improving bone density.

Post-operative Evaluation Post-surgery, patients receive instructions and medications for post-operative care. A follow-up DentaScan CT is performed to assess changes in bone density at the implant sites, comparing these post-operative measurements to the pre-operative baselines to evaluate the effectiveness of the osseodensification technique.

Data Analysis Data from pre-operative and post-operative evaluations are systematically recorded and analyzed using SPSS software. A student paired t-test is utilized to ascertain the significance of changes in bone density, with a p-value of less than 0.05 deemed statistically significant.

Objective The primary aim is to ascertain whether the use of osseodensification drilling techniques yields a measurable improvement in bone density around implant sites, potentially enhancing dental implant success rates by fostering better primary stability and facilitating osseointegration.

Significance The study seeks to offer empirical evidence supporting the application of osseodensification in dental implantology. By rigorously assessing the technique's impact on bone density and implant stability, the research endeavors to make a meaningful contribution to surgical practices in dental implant placement, aiming to ultimately enhance patient outcomes by leveraging this innovative technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partial or complete edentulous ridge in the maxilla or mandible.

Exclusion Criteria:

* Presence of a fractured jaw.
* General bone or blood disorders that may affect osseointegration

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase in Bone Density at Implant Sites Using Osseodensification Technique | 3-6 months
  The primary outcome measure is the change in bone density at the dental implant sites, measured in Hounsfield units (HU), from pre-operative to post-operative stages. The study aims to quantify the effectiveness of the osseodensification technique in enhancing bone density around the implant sites, thereby potentially improving the primary stability of dental implants. The outcome will be assessed using DentaScan CT imaging analyzed with Radiant DICOM software to compare bone density values at apical, mesial, and distal positions relative to each implant site before and after the surgical intervention.

IPD SHARING:
Plan to Share IPD: No
The study aims to share specific individual participant data related to the osseodensification technique's effect on bone density around dental implant sites. Data to be shared includes pre-operative and post-operative bone density measurements at specified implant sites, measured in Hounsfield units, and statistical analyses comparing these measurements. The data will be anonymized to protect participant confidentiality and shared with researchers who provide a methodologically sound proposal for purposes of advancing knowledge in dental implant stability and bone density impacts. Data will be available upon request following publication of the study results, subject to approval by the study's ethical review board and under a data-sharing agreement that specifies data use, security requirements, and data destruction upon project completion.

REFERENCES:
- [Derived] Vaddamanu SK, Saini RS, Vyas R, Kanji MA, Alshadidi AAF, Hafedh S, Cicciu M, Minervini G. A comparative study on bone density before and after implant placement using osseodensification technique: a clinical evaluation. Int J Implant Dent. 2024 Nov 19;10(1):56. doi: 10.1186/s40729-024-00565-8. PMID 39560860